CLINICAL TRIAL: NCT01213576
Title: Efficacy of Higher Albendazole and Ivermectin Doses on Wuchereria Bancrofti Microfilarial Clearance in Malawi, Open Label Study
Brief Title: Efficacy of Higher Albendazole and Ivermectin Doses on Wuchereria Bancrofti Microfilarial Clearance in Malawi
Acronym: FED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Introduction of National Mass Drug Administration Campaign and failure to identify appropriate participants.
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Neil French, Reader In Infectious Disease Epidemiology/Director KPS, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FED-311207
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Lymphatic Filariasis
Keywords: Lymphatic filariasis; microfilaria; Albendazole; ivermectin; human immunodeficiency
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- albendazole 400mg and ivermectin 200mcg/kg (Active Comparator): Annual treatment
  Interventions: Drug: Albendazole 400mg and ivermectin 200mcg/kg
- Albendazole 800mg and ivermectin 400mcg/kg (Active Comparator): Annual treatment
  Interventions: Drug: Albendazole and ivermectin
- Albendazole 400mg and ivermectin 200mcg/kg (Active Comparator): albendazole 400mg and ivermectin 200mcg/kg given twice a year
  Interventions: Drug: Albendazole 400mg and ivermectin 200mcg/kg
- Albendazole 800mg and ivermectin 400mcg /kg bi-annually (Active Comparator): Albendazole 800mg and ivermectin 400mcg/kg given twice a year
  Interventions: Drug: albendazole 800mg and ivermectin 400mcg/kg bi-annually

INTERVENTIONS:
Drug: Albendazole 400mg and ivermectin 200mcg/kg — 400 mg orally given annually
  Arms: Albendazole 400mg and ivermectin 200mcg/kg; albendazole 400mg and ivermectin 200mcg/kg
Drug: Albendazole and ivermectin — albendazole 800 mg and ivermectin 400mg orally given annually
  Arms: Albendazole 800mg and ivermectin 400mcg/kg
Drug: Albendazole 400mg and ivermectin 200mcg/kg — Albendazole 400mg and ivermectin 200mcg/kg given twice a year
  Arms: Albendazole 400mg and ivermectin 200mcg/kg; albendazole 400mg and ivermectin 200mcg/kg
Drug: albendazole 800mg and ivermectin 400mcg/kg bi-annually — albendazole 800mg and ivermectin 400mcg/kg given twice a year
  Arms: Albendazole 800mg and ivermectin 400mcg /kg bi-annually

SUMMARY:
Albendazole and ivermectin are currently used in combination for annual mass treatment of lymphatic filariasis in Africa. Although the drugs have been donated, the cost of such programmes is very high and has proven to be a major impediment to the success of programmes in many countries with limited financial resources.

Data from albendazole treatment of other filarial infections and one study comparing single to multi-dose Diethycarbamazine/albendazole in lymphatic filariasis suggest that increased dose and/or frequency of albendazole dosing may be more effective in clearing microfilariae. It is essential to determine whether such higher doses are indeed beneficial since this could have far-reaching effects on the conduct and management of the main mass treatment programmes and also in the management of programmes as they near elimination.

DETAILED DESCRIPTION:
The proposed study will enrol up to 120 volunteers with microfilaremic Wuchereria bancrofti infection who would be randomized to receive standard annual treatment (albendazole 400 mg + ivermectin 200 mcg/kg), annual treatment with an increased dose of albendazole (albendazole 800 mg + ivermectin 200400 mcg/kg) or semi-annual treatment with a standard (albendazole 400 mg + ivermectin 200 mcg/kg), or an increased albendazole dose (albendazole 800 mg + ivermectin 200 400 mcg/kg). Microfilarial levels, as well as measures of adult worm burden (circulating antigen) will be followed every six months for two years to determine whether the higher doses, or more frequent regimens are more effective.

The data obtained would be used, in combination with the data from other similar studies being conducted in Mali and in India to advise the Global Programme for the Elimination of Lymphatic Filariasis (GPELF) on improved methods of treatment both for mass treatment and for the management of problem areas within the global programme.

ELIGIBILITY:
Inclusion Criteria:

* understand and sign informed consent
* willing to undergo night blood sampling every 6 months for 2 years
* Age 18 to 55 years
* Haemoglobin of equal or above 9g/dl
* Microfilarial level of equal or above 80mg/dl

Exclusion Criteria:

* Non- consenting
* Pregnancy or lactation
* Treatment with albendazole or ivermectin within the previous 6 months
* Known allergy to the study drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil French, MB ChB PHD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Karonga Prevention Study, Karonga, Malawi

REFERENCES:
- [Derived] Tafatatha TT, Ngwira BM, Taegtmeyer M, Phiri AJ, Wilson TP, Banda LG, Piston WN, Koole O, Horton J, French N. Randomised controlled clinical trial of increased dose and frequency of albendazole and ivermectin on Wuchereria bancrofti microfilarial clearance in northern Malawi. Trans R Soc Trop Med Hyg. 2015 Jun;109(6):393-9. doi: 10.1093/trstmh/trv027. Epub 2015 Apr 15. PMID 25877874

RESULTS

PARTICIPANT FLOW:
Groups:
- Albendazole 400mg and Ivermectin 200mcg/kg Annually: Once a year treatment
  Albendazole 400mg and ivermectin 200mcg/kg: 400 mg oral
- Albendazole 800mg and Ivermectin 400mcg/kg Annually: Once a year treatment
  Albendazole and ivermectin: albendazole 800 mg and ivermectin 400mg oral
- Albendazole 400mg and Ivermectin 200mcg/kg Biannually: Twice a year
  albendazole 400mg and ivermectin 200mcg/kg given twice a year
- Albendazole 800mg and Ivermectin 400mcg /kg Bi-annually: Twice a year
  Albendazole 800mg and ivermectin 400mcg/kg given twice a year
Period: Overall Study
Arm/Group | Albendazole 400mg and Ivermectin 200mcg/kg Annually | Albendazole 800mg and Ivermectin 400mcg/kg Annually | Albendazole 400mg and Ivermectin 200mcg/kg Biannually | Albendazole 800mg and Ivermectin 400mcg /kg Bi-annually
Started | 18 | 17 | 18 | 17
Completed | 15 | 13 | 13 | 13
Not Completed | 3 | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Albendazole 400mg and Ivermectin 200mcg/kg Annual: Albendazole 400mg and ivermectin 200mcg/kg: 400 mg orally given once a year
- Albendazole 800mg and Ivermectin 400mcg/kg Annual: Albendazole and ivermectin: albendazole 800 mg and ivermectin 400mg orally given once a year
- Albendazole 400mg and Ivermectin 200mcg/kg Biannual: Albendazole 400mg and ivermectin 200mcg/kg given twice a year
- Albendazole 800mg and Ivermectin 400mcg/kg Bi-annual: Albendazole 800mg and ivermectin 400mcg/kg given twice a year
- Total: Total of all reporting groups
Arm/Group | Albendazole 400mg and Ivermectin 200mcg/kg Annual | Albendazole 800mg and Ivermectin 400mcg/kg Annual | Albendazole 400mg and Ivermectin 200mcg/kg Biannual | Albendazole 800mg and Ivermectin 400mcg/kg Bi-annual | Total
Number analyzed (Participants) | 18 | 17 | 18 | 17 | 70
Age, Continuous [Median (Full Range); unit: years] | 32.5 [21 to 50] | 31 [20 to 53] | 27.5 [18 to 55] | 35 [20 to 54] | 33 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 7 | 7 | 23
  Male | 15 | 11 | 11 | 10 | 47
Region of Enrollment [Number; unit: participants]
  Malawi | 18 | 17 | 18 | 17 | 70
Microfilarial count /uL [Geometric Mean (Full Range); unit: microfilaria/uL] | 464.7 [250.1 to 863.4] | 338.7 [198.7 to 577.4] | 204.5 [204.5 to 287.8] | 264.7 [175.0 to 400.4] | 298.6 [207.3 to 389.4]
HIV status [Number; unit: participants] | 0 | 0 | 0 | 0 | 0
Eosinophil count [Geometric Mean (Full Range); unit: cells/uL] | 1300 [1000 to 1700] | 1400 [1000 to 1900] | 1600 [1100 to 2100] | 1100 [900 to 1500] | 1300 [1000 to 1800]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Microfilarial Clearance
Description: Microfilaria clearance will be assessed in regard to dosage as well as frequency of treatment. Microfilarial clearance is defined by non-detection of microfilaria in the night blood sample.
Time Frame: 12 months
Population: Number of participants with non detectable microfilaria at follow up
Measure: Number; unit: participants
Arm/Group | Albendazole 400mg and Ivermectin 200mcg/kg Annually | Albendazole 800mg and Ivermectin 400mcg/kg Annually | Albendazole 400mg and Ivermectin 200mcg/kg Biannually | Albendazole 800mg and Ivermectin 400mcg /kg Bi-annually
Number analyzed (Participants) | 18 | 17 | 18 | 17
participants | 15 | 14 | 13 | 17

2. Secondary Outcome: Number of Participants With Microfilarial Clearance at 24 Months of Follow up
Description: Microfilaria will be detected using the nucleopore filtration technique and analysed according to the respective treatment arms at the 24 month time point. Microfilarial clearance will be defined by non-detection of microfilaria in the night blood sample
Time Frame: 24 months
Population: Intention to treat, with last result carried forward in the case of missing visit
Measure: Number; unit: participants
Arm/Group | Albendazole 400mg and Ivermectin 200mcg/kg Annually | Albendazole 800mg and Ivermectin 400mcg/kg Annually | Albendazole 400mg and Ivermectin 200mcg/kg Biannually | Albendazole 800mg and Ivermectin 400mcg /kg Bi-annually
Number analyzed (Participants) | 18 | 17 | 18 | 17
participants | 17 | 17 | 14 | 17

ADVERSE EVENTS:
Arm/Group | Albendazole 400mg and Ivermectin 200mcg/kg Annually | Albendazole 800mg and Ivermectin 400mcg/kg Annually | Albendazole 400mg and Ivermectin 200mcg/kg Biannually | Albendazole 800mg and Ivermectin 400mcg /kg Bi-annually
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 5/18 | 7/17 | 6/18 | 4/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albendazole 400mg and Ivermectin 200mcg/kg Annually (N=18) | Albendazole 800mg and Ivermectin 400mcg/kg Annually (N=17) | Albendazole 400mg and Ivermectin 200mcg/kg Biannually (N=18) | Albendazole 800mg and Ivermectin 400mcg /kg Bi-annually (N=17)
Fever (General disorders) | 2 | 4 | 3 | 1
headache (General disorders) | 3 | 4 | 4 | 2
joint pains (General disorders) | 2 | 1 | 3 | 2
abdominal pains (General disorders) | 1 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes